CLINICAL TRIAL: NCT00369837
Title: Evaluation of the Effect of Ultrashort-Acting Clevidipine in the Treatment of Patients With Severe Hypertension (VELOCITY)
Brief Title: Clevidipine in the Treatment of Patients With Severe Hypertension (VELOCITY)
Acronym: VELOCITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMC-CLV-06-02; VELOCITY (Other: Sponsor)
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — clevidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- clevidipine (Experimental): A patient-specific blood pressure target range (TR) of ≥20 mm Hg and ≤40 mm Hg SBP was prespecified by the investigator. Once established, clevidipine (0.5 mg/mL in 20% lipid emulsion) intravenous infusion was initiated at 2.0 mg/h and maintained for the first 3 minutes. Clevidipine was up-titrated, as tolerated by the patient, by doubling the dose every 3 minutes until the prespecified systolic blood pressure (SBP) target range was achieved and could continue to be titrated up or down to maintain the desired long-term SBP reduction.
  Interventions: Drug: clevidipine

INTERVENTIONS:
Drug: clevidipine — Clevidipine was required to be administered continuously for a minimum of 18 hours and a maximum of 96 hours and was not to exceed a rate of 32.0 mg/h at any time. Use of an additional or alternative intravenous antihypertensive agent was allowed if the blood pressure target range was not achieved or maintained. If transition to an oral antihypertensive agent is required, then approximately 1 hour prior to the anticipated cessation of clevidipine infusion, but no less than at the 18-hour time point, an oral antihypertensive agent was allowed to be administered as clevidipine was down-titrated or terminated as needed in order to achieve the desired blood pressure level..
  Other Names: clevidipine, Cleviprex

SUMMARY:
The purpose of this study was to determine the safety of clevidipine for treating severely elevated blood pressure, defined as systolic (SBP) >180 mmHg and/or diastolic blood pressure (DBP) >115 mmHg assessed on 2 successive occasions 15 minutes apart at baseline, in patients with or without major organ injury, particularly with respect to controlled dose adjustment to desired effect and prolonged continuous infusion. Enrollment of patients into the study was to continue until the target goal of 100 patients with at least 18 hours of continuous clevidipine treatment, including a minimum of 50 patients with acute or chronic end-organ injury, was met.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Systolic blood pressure >180 mmHg and/or diastolic blood pressure >115 mmHg assessed on two successive occasions, 15 minutes apart at baseline
* Written informed consent

Exclusion Criteria:

* SBP ≤180 mmHg and/or DBP ≤115 mmHg
* Expectation that the patient will not tolerate intravenous antihypertensive therapy for at least 18 hours
* Known or suspected aortic dissection
* Administration of an agent for treating hypertension within 2 hours of clevidipine administration
* Severe hypertension known to be precipitated by use of, or withdrawal from, alcohol or illicit drugs, or intentional overdose of illicit or prescription drugs
* Positive pregnancy test
* Intolerance to calcium channel blockers
* Allergy to soybean oil or egg lecithin
* Known liver failure or cirrhosis
* Participation in clinical research studies of other investigational drugs or devices within 30 days of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2006-09; Primary Completion 2007-01 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients in whom SBP falls below the lower limit of the patient-specific, pre-determined blood pressure target range at the initial dose (2.0 mg/h) | Study drug initiation through the first 3 minutes of the infusion
Percentage of patients who reach the prespecified target SBP range | Within 30 minutes of the initiation of the infusion

SECONDARY OUTCOMES:
Time to attainment of the 30-minute SBP target range | During the 30-minute period from initiation of infusion
Change in heart rate | During the 30-minute period from initiation of infusion
Mean and median dose of clevidipine during the treatment period | Treatment period is from initiation of infusion until study drug termination (minimum of 18 hours up to a maximum of 96 hours)
Proportion of patients transitioning to oral antihypertensive therapy | Within 6 hours of stopping study drug infusion
Safety of clevidipine infusion for 18 hours or longer | Treatment period is from initiation of infusion until study drug termination (minimum of 18 hours up to a maximum of 96 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Charles V Pollack, MA MD FACEP, Principal Investigator — Pennsylvania Hospital; Frank Peacock, MD FACEP, Principal Investigator — The Cleveland Clinic
Locations (14):
- United States (14):
  - Jackson Hospital, Montgomery, Alabama
  - VA Medical Center W. LA, Los Angeles, California
  - The George Washington University Medical Center, Washington D.C., District of Columbia
  - Louisiana State University Medical Center/Charity Hospital, New Orleans, Louisiana
  - Critical Care Research Center at Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Good Samaritan Hospital, Baltimore, Maryland
  - Duke University Medical Center, Durham, North Carolina
  - Metrohealth Medical Center, Cleveland, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Providence Heart & Vascular Institute, d/b/a Providence St. Vincent Medical Center, Portland, Oregon
  - Hamot Shock Trauma, Erie, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - The University of Texas Health Science Center, Houston, Texas

REFERENCES:
- [Result] Pollack CV, Varon J, Garrison NA, Ebrahimi R, Dunbar L, Peacock WF 4th. Clevidipine, an intravenous dihydropyridine calcium channel blocker, is safe and effective for the treatment of patients with acute severe hypertension. Ann Emerg Med. 2009 Mar;53(3):329-38. doi: 10.1016/j.annemergmed.2008.04.025. Epub 2008 Jun 5. PMID 18534716